CLINICAL TRIAL: NCT00243282
Title: Randomized Controlled Trial of Mind-Body Breathing Therapy (in Chronic Obstructive Pulmonary Disease) To Improve Palliation of Dyspnea and Health-Related Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Samueli Institute for Information Biology (Other)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S05-Shekelle0024; PCC 2005-081225
Record Dates: First submitted 2005-10-19; First posted 2005-10-21 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2008-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Complementary Therapies; Dyspnea; Palliative Care; Meditation; Quality of Life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): Control (Support Group)
- 2 (Other): Intervention (Mindfulness Based Breathing Therapy)
  Interventions: Behavioral: Relaxation Response (instruction, pocket practice card prov); Behavioral: Mindfulness training using model developed from UMass

INTERVENTIONS:
Behavioral: Relaxation Response (instruction, pocket practice card prov)
  Arms: 2
Behavioral: Mindfulness training using model developed from UMass
  Arms: 2

SUMMARY:
Dyspnea (shortness of breath) is a complex experience that includes interpretation of physical impairments and associated distress to the person. The role of mind-body interactions in the experience of the symptom of dyspnea suggests that complementary and alternative medicine (CAM) therapies may be effective in abating dyspnea and improving patients' health-related quality of life. CAM strategies work in a number of ways that are directly applicable to dyspnea, such as decreasing the stress response, inducing relaxation, and facilitating a less distressful interpreted experience of physical disorders.

We have combined a number of established CAM approaches aimed at breath-centered mindfulness and relaxation into an single therapy, mind-body breathing therapy (MBBT). The purpose of this study is to test the efficacy of MBBT in improving dyspnea and health-related quality of life for patients with emphysema (chronic obstructive pulmonary disease).

DETAILED DESCRIPTION:
Objectives We aim to test the feasibility and efficacy of mind-body breathing therapy (MBBT) in improving dyspnea and health-related quality of life for patients suffering from late-stage COPD. This randomized controlled trial seeks to assimilate a number of complementary and alternative (CAM) approaches aimed at breath-centered symptom abatement and relaxation into an single therapy and test its efficacy as a palliative care intervention.

Research Plan Patients will be enrolled from outpatient clinics, primarily pulmonary medicine (COPD patients), at the Veteran Affairs (VA) Greater Los Angeles Healthcare System. Patients will be randomized to intervention or control arms. Each arm will include a weekly meeting on the VA campus for 8 successive weeks. Evaluation will include pre/post measurements, serial self-report data, compliance measures, chart abstracted objective data, and follow-up evaluations for 2 months following the intervention or until death. Grant and project will begin in October 2005 and run for one year.

Methods The overall design is a randomized controlled trial of the MBBT intervention on dyspnea symptoms and health-related quality of life (HRQOL). The study will aim to enroll 120 patients over a one year period. We will enroll cognitively intact patients with advanced COPD and dyspnea. Potential subjects will be identified by flyers or provider invitation; screening will ask about enrollment criteria and verified after consent through medical record. Subjects will be recruited through physicians though public advertising and recruitment within the VA will be used to inform patients and physicians of the trial. Patients will be screened at intake during vital signs and offered participation when identified with dyspnea of at least 4 out of 10 points on the Borg Dyspnea Scale. Patients randomized to intervention arm will attend a 8-week session on MBBT that will include a 15 minute video designed by Jon Kabat-Zinn for dyspnea, a relaxation response pocket-guide with group practice and a daily prescription for practice, and weekly mind-body guided sessions for controlled breathing. Control patients will be invited to attend an 8-week session consisting of the a support group with equivalent time and attention as well as identical measures.

Results Primary study outcomes are patients' self report of the severity of dyspnea and HRQOL. Baseline dyspnea will be quantified with the Baseline Dyspnea Index and Borg scale with regular measures of dyspnea using the Visual Analog Scale (VAS). Functional limitation will be measured by the 6-minute walk test and followed with the baseline measure of post-exercise dyspnea level on the Borg scale. Other symptoms will be identified by the Memorial Symptom Assessment Scale (MSAS) and as part of the Saint George Respiratory Questionnaire (SGRQ). HRQOL will be measured by the SGRQ, a 76-item self-administered questionnaire measuring 3 domains (symptoms, activity, and impact of disease on daily life), and in a more general way by the physical health score and mental health score of the Veterans RAND 36 Item Health Survey (VR-36).

Clinical Significance Chronic obstructive pulmonary disease (COPD) is the fourth leading cause of death with increasing prevalence throughout the world and within the VA. Dyspnea is among the most troublesome symptoms these patients experience. Mindfulness based meditative strategies has been shown to improve functioning and quality of life, and palliate pain in other populations. However, no trial has specifically evaluated mindful practices or mind-body breathing techniques in the palliation of dyspnea. If shown to be effective, MBBT may represent an important palliative strategy in the management of conditions prevalent in the Veteran population and in medical care in general.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Obstructive Pulmonary Disease
* Resting Dyspnea > 2 OR Activity Dyspnea > 4 in the prior 4 weeks to screening

Exclusion Criteria:

* Cognitive impairment on the 10-item Short Portable Mental Status Questionnaire
* History of serious psychiatric illness
* Unwilling or unable to participate in the full eight week program and evaluation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120
Dates: Start 2005-10; Study Completion 2006-10

PRIMARY OUTCOMES:
Primary study outcomes are patients' self report of the severity of dyspnea and HRQOL. Baseline dyspnea will be quantified with the Baseline Dyspnea Index and Borg scale with regular measures of dyspnea using the Visual Analog Scale (VAS). HRQOL will be | 8 weeks

SECONDARY OUTCOMES:
Functional limitation will be measured by the 6-minute walk test and followed with the baseline measure of post-exercise dyspnea level on the Borg scale. Other symptoms will be identified by the Memorial Symptom Assessment Scale (MSAS) and as part of the | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul G. Shekelle, MD, PhD, Principal Investigator — Greater Los Angeles VA Healthcare System, Chief General Internal Medicine
Locations (1):
- Greater Los Angeles VA Healthcare System, Los Angeles, California, United States

REFERENCES:
- [Derived] Mularski RA, Munjas BA, Lorenz KA, Sun S, Robertson SJ, Schmelzer W, Kim AC, Shekelle PG. Randomized controlled trial of mindfulness-based therapy for dyspnea in chronic obstructive lung disease. J Altern Complement Med. 2009 Oct;15(10):1083-90. doi: 10.1089/acm.2009.0037. PMID 19848546